CLINICAL TRIAL: NCT03555773
Title: Treatment of Complex Crohns' Perianal Fistulas by Local Injection of Autologous and Micro-fragmented Adipose Tissue
Brief Title: Micro-fragmented Adipose Tissue and Complex Crohns' Anal Fistulas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Silvio Laureti, Associated Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lipogems-crohn2
Record Dates: First submitted 2018-05-22; First posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Crohn Disease; Perianal Fistula
Keywords: perianal Crohn's disease; mesenchymal stromal cells; complex anal fistulas; micro-fragmented adipose tissue; regenerative medicine
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: 15 patients with complex fistulizing perianal Crohn's disease refractory to biological therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lipogems (Experimental): Lipogems injection into the submucosa surrounding the internal fistula orifice and in the perianal tissue along the residual fistula tract
  Interventions: Procedure: Lipogems

INTERVENTIONS:
Procedure: Lipogems — After local surgical drainage of the perianal disease, micro-fragmented adipose tissue is injected circumferentially into the submucosa surrounding the internal fistula orifice and in the perianal tissue along the residual fistula tract.

SUMMARY:
The study aims to evaluate safety, feasibility and effectiveness of local injections of autologous and micro-fragmented adipose tissue obtained with the Lipogems® system in patients with refractory complex fistulizing perianal Crohn's disease.

DETAILED DESCRIPTION:
Complex perianal fistulas represent one of the most challenging manifestations of Crohn's disease. Combined surgical and medical therapy with biologic drugs today represents the first-line treatment option but the overall success rate does not exceed 60%. The treatment of patients in which complete closure cannot be achieved despite the combination of biological therapy and surgery, is still not well defined. These patients may benefit from innovative therapeutic approaches such as mesenchymal stromal cells. The adipose tissue is an ideal source, due to its abundance and easy access. The investigators evaluate safety, feasibility and effectiveness of local injections of micro-fragmented adipose tissue in patients with refractory complex fistulizing perianal Crohn's disease.

STUDY DESIGN This is a no profit interventional prospective study without drugs. A cohort of patients (15) with complex perianal Crohn's Disease, refractory to standard treatment with biologic drugs, or with secondary failure after initial effectiveness or presenting clinical contraindications to biological treatment are enrolled in the study.

After the enrolment, medical history and clinical data are collected and pre-operatory exams, pelvic MRI, and laboratory tests (erythrocyte sedimentation rate and C-reactive protein) are performed. Health-related quality of life is assessed by a disease-specific (Inflammatory Bowel Disease Questionnaire) and a generic (Short-Form 36 Health Survey) questionnaire.

METHODS

- Harvesting of the adipose tissue

The lower/lateral abdomen or, eventually, the inner/outer thigh are chosen as donor site for adipose tissue harvesting under general or spinal anaesthesia. Before the harvesting, the donor site is injected with 100 cc of Klein Solution (500 cc saline, 1 cc epinephrine 1/1000 IU, and 40 cc lidocaine 2%) using a disposable 17 gauge blunt cannula connected to a 60-cc luer-lock syringe. The fat is then harvested (50-100 cc) using a 13 gauge blunt cannula connected to a 20-ml VacLok® syringe.

- Processing of the adipose tissue with the Lipogems® device

The harvested fat is immediately processed in the Lipogems® processing kit (Lipogems International Spa, Milan, Italy). Lipogems® is a disposable device that mechanically reduces the size of the adipose tissue clusters while eliminating oily substances and blood residues with pro-inflammatory properties. The entire process is carried out in one surgical step in complete immersion in physiological solution minimizing any traumatic action on the cells and microarchitecture. The processed micro-fragmented fat is collected in a 60-cc syringe and positioned to decant the excess of saline solution. At the end, the product is transferred in several 5-cc syringes to be re-injected in the patient.

- Surgical procedure and micro-fragmented adipose tissue (Lipogems®) injection

Examination under anaesthesia is performed in order to identify all the fistula tracts and abscesses; eventual purulent material is drained and the fistula tracts curetted. Necrotic and inflamed tissues are excised using a "cone-like" fistulectomy at each fistula tract. After local surgical drainage of the perianal disease, 20 cc of micro-fragmented adipose tissue are injected circumferentially into the submucosa surrounding the internal fistula orifice and in the perianal tissue along the residual fistula tract.

- Follow-up visits and outcome measures

All patients are assessed at 2, 4, 8, 12 and 24 weeks after the procedure. During all follow-up visits, laboratory tests and clinical examination are performed. health related quality of life questionnaires are also administered. A second pelvic MRI is performed at 24 weeks to radiologically assess the results.

ELIGIBILITY:
Inclusion Criteria:

* Signature of the informed consent
* Diagnosis of Crohn's Disease confirmed by instrumental and histological methods
* Age >18 years; both genders
* Presence of complex fistulizing perianal Crohn's Disease refractory to standard treatment (combination of surgical drainage of sepsis and local/systemic administration of anti-tumor necrosis factor-alpha agents with subsequent surgical "rescue" repair by means of endoanal mucosal flap or biological plug placement).

Exclusion Criteria:

* Patients unable to follow the schedule of the protocol
* Patients with ano- and recto-vaginal fistulas
* Patients with active infections by Human Immunodeficiency Virus, hepatitis C virus, hepatitis B virus, tuberculosis, septic uncontrolled conditions
* Patients with abdominal acute localization of Crohn's Disease that could have required general surgery during the study
* Patients with oncological or lymphoproliferative active diseases
* Patients where an adequate amount of lipoaspirate (at least 60 cc) could not be safely harvested

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
Healing | 6 months
  Closing of the fistula tract clinically assessed and confirmed by pelvic MRI

SECONDARY OUTCOMES:
Health-related quality of life assessed by a disease specific questionnaire | 6 months
  Health-related quality of life assessed by changes from baseline evaluation to 6 months follow-up of the Inflammatory Bowel Disease Questionnaire (IBDQ). The questionnaire is made of 32 questions grouped into four dimensions: bowel, systemic, social, and emotional. Scores range from 1 (denoting a very severe problem) to 7 (denoting no problem at all). Scale range: worst quality of life: 32 - best quality of life: 224. Meaningful change is estimated at 16 points for the overall score.
Health-related quality of life assessed by a generic questionnaire | 6 months
  Health-related quality of life assessed by changes from baseline evaluation to 6 months follow-up of the Short-Form 36 Health Survey (SF-36) questionnaire.
  The SF-36 is a generic questionnaire with 36 items that measure functional health and well-being. It comprises eight domains and two psychometrically-established summary components, each derived from four domain scores. Domain and summary component scores range from 0-100; higher scores correspond to better health status or well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto Poggioli, Prof, Principal Investigator — S. Orsola-Malpighi Hospital, Department of Medical and Surgical Sciences (DIMEC), University of Bologna, Bologna
Locations (1):
- S. Orsola-Malpighi Hospital, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided